CLINICAL TRIAL: NCT07180732
Title: Accuracy of Direct Composite Veneers Using Injection Moulding Technique
Brief Title: Accuracy of Injection Moulding Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NewGiza University (Other)
Responsible Party: Principal Investigator, Omar Shaalan, Associate professor of conservative dentistry, NewGiza University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Accuracy of injection mouldong
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Esthetic Restorations
Keywords: Injection moulding; Veneers; Accuracy; Geomagic; resin composite

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injection moudling technique (Experimental): A dental procedure where a patient-approved tooth shape, established from a diagnostic wax-up, is replicated using a transparent silicone index
  Interventions: Procedure: Injection moulding technique
- Digital smile design (Other): Baseline smile design
  Interventions: Diagnostic Test: Digital smile design

INTERVENTIONS:
Procedure: Injection moulding technique — A dental technique that uses a transparent silicone index or stent to inject a low-viscosity composite into a pre-planned and approved tooth shape.
  Arms: Injection moudling technique
Diagnostic Test: Digital smile design — A modern approach that uses digital imaging, videos, and software to create a customized, virtual 3D model of a patient's ideal smile before any treatment begins
  Arms: Digital smile design

SUMMARY:
To evaluate the discrepancy between the digital smile design (DSD) and the resulting direct composite veneers via Injection Moulding Technique.

DETAILED DESCRIPTION:
This study will be aiming at testing the accuracy of the injection moulding technique compared with the digital smile design, therefore improving the outcome of composite veneers for the patients in order to reach more predictable results. Utilizing a quantitative method to assess accuracy of Injection moulding technique is deficient in literature and using a geometrical subtraction software will be an objective method to compare the difference with the digital smile design.

ELIGIBILITY:
Inclusion Criteria:

* Participants requiring smile make-over
* Good oral hygiene
* Compliance

Exclusion Criteria:

* Poor oral hygiene
* Need for orthodontic treatment
* Need of full coverage restoration
* Parafunctional habits
* Lack of compliance

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Accuracy | From enrolment to the end of treatment after 4 weeks
  The root mean square (RMS) values were obtained through the "3D-compare" method followed by comparison at each surface point between the reference digital design desing and the final outcome using injection moulding

CONTACTS AND LOCATIONS:
Overall Officials: Omar O Shaalan, PhD, Principal Investigator — Associate Professor, Department of conservative dentistry
Locations (1):
- School of dentistry, Newgiza University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to concerns regarding participant privacy and the absence of explicit consent for data sharing